CLINICAL TRIAL: NCT06531902
Title: LncRNA NNT-AS1/Hsa-miR-485-5p/HSP90 Axis In-silico and Clinical Prospect correlated-to Histologic Grades-based CRC Stratification: A Step Toward ncRNA Precision
Brief Title: LncRNA Nicotinamide Nucleotide Transhydrogenase-Antisense RNA1 NNT-AS1 in CRC
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Prof. Nadia M. Hamdy, Ph.D., professor of biochemistry and molecular biology, Ain Shams University
Other Study IDs: REC #293
Record Dates: First submitted 2024-05-16; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; LncRNA NNT-AS1; Hsa-miR-485-5p; HSP90; Prognositic molecular biomarkers
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Five milliliters of peripheral venous blood liquid biopsy were collected from the antecubital vein from controls and CRC patients into clot activator polymer gel vacutainers (Greiner Bio-One GmbH, Australia). Vacutainers of completely coagulated samples were centrifuged at 4000 r.p.m for 10 min at room temperature (25 ◦C). The collected serum was aliquoted and kept at - 80 ◦C in three DNase/ RNase free Eppendorf tubes until analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: A total of 60 CRC pateints' were enrolled in the study. CRC pateints' were treatment-naïve Egyptian patients' cohort admitted to the Clinical Oncology Clinic, National Cancer Institute (NCI), Cairo University, Cairo, Egypt. Male-to-female 1:1 (30/30) and their age range 24-76 years.
- Healthy Control: 28 age-matched and sex-matched apparently healthy volunteers, randomly selected from subjects enlisted during normal check-up examination or during blood donation. The control group participants were not taking any medication or suffering from any disease. Controls age range is 40-60 years and 13:15 male-to-female.

SUMMARY:
The current study will compare the blood expression level of lncRNA NNT-AS1 and hsa-miR-485-5p, as well as heat shock protein 90 (HSP90) serum levels in both healthy and CRC Egyptian patients' cohort peripheral blood samples. Second, examine if lncRNA NNT-AS1/hsa-miR-485 5p/HSP90 axis, or individually investigated, would be used as a non-invasive molecular precision biomarker in liquid biopsy for better diagnostic utility for CRC patients. Also, based on CRC patients' group stratification by histologic grades 1-3. Finally, investigate the probable link/correlation between lncRNA NNT-AS1/hsa-miR-485-5p/HSP90 as an axis or individually in CRC Egyptian patients' cohort in relation to demographic data or clinicopathological characteristics. All findings will be confirmed or ruled out by in silico means as well.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a heterogeneous malignancy that affects the colon and rectum. It is the third most prevalent and lethal malignancy, with roughly 1.9 million new cases and nearly 9.4% of cancer-related deaths in 2020 worldwide. The CRC survival rate mostly relies on the disease's stage at the time of diagnosis. Thus, early detection of CRC provides a higher 5-year survival probability of 80-90%, compared to just 14% in the late stage with distant metastases. Colonoscopy is the gold standard method for CRC diagnosis. Alongside its great accuracy, it is an invasive technique with considerable mortality risks, such as intestinal perforation and bleeding, limiting its usage for screening. Fecal occult blood test, carbohydrate antigen 19-9 (CA19-9) and carcinoembryonic antigen (CEA) are the currently available CRC early diagnosis screening/ tumor markers (TMs) tests. Although CEA and CA19-9 tests are simple, non-invasive, affordable, and safe, their diagnostic accuracy is limited. Screening and early diagnosis for CRC have been identified as the most significant factor for lowering mortality. Long non-coding RNA (lncRNA), which are more than 200 nucleotides non-coding RNAs (ncRNAs), are either over-expressed or down-regulated in numerous malignancies, and act as potential molecular mediators for various tumors progression. Overexpressed lncRNAs act as oncogenes enhancing tumor cell proliferation, apoptosis, invasion, metastasis, and autophagy. Several lncRNAs have been linked to the incidence, metastasis, and therapeutic resistance of CRC. Recent research suggested that the lncRNA Nicotinamide Nucleotide Transhydrogenase-antisense RNA1 (NNT-AS1), which is localized in the 5p12 human chromosome, is involved in gene expression regulation and plays important roles in a variety of cancers, such as breast cancer, cervical cancer, hepatocellular carcinoma, and osteosarcoma, however, insufficient research was performed about lncRNA NNT-AS1 role in CRC. MicroRNAs (miRNAs) are small ncRNAs with ~22 nucleotides length, that undertake a variety of biological functions such as cell proliferation, apoptosis, and angiogenesis. The mature miRNA species, also known as the miRNA-5p (guide' strand) and - 3p species (passenger miRNA), can originate from both the 5' and 3' arms of the precursor duplex. The arm that is destined to be loaded into the RNA-induced silencing complex is the guide strand. Passenger miRNAs were assumed to be entirely destroyed, however, deep sequencing investigations have revealed that certain minor miRNAs retain and, in fact, play a meaningful role in gene regulation. Numerous studies have found a substantial association between miRs dysregulation and tumor metastasis. Homo sapiens (hsa)-miR-485-5p is located on the human chromosome 14q32 and has been identified as an anticancer/tumor suppressor gene in several human malignancies, through targeting and regulating the expression of downstream cell proliferation and invasion genes. The regulatory function of hsa-miR-485-5p in CRC is still undetermined. LncRNAs-miRs interaction would control the incidence and/or progression of various cancer types, as well as being considered as potential target for future treatment invention. LncRNA NNT-AS1 was found to promote proliferation, migration, and invasion of cholangiocarcinoma via sponging hsa-miR-485. This sponging process elevated β-catenin and B-cell chronic lymphocytic leukemia (CLL)/lymphoma 9 (BCL9) in response. LncRNA NNT-AS1's relation to hsa-miR-485-5p in CRC remains to be determined clinically. In most cells, under non-stress settings, heat shock protein 90 (HSP90) are highly conserved molecular chaperones that make up 1-2% of all cellular proteins. Important functions of HSP90 proteins include protein folding and degradation. Physiologically, the molecular chaperone HSP90AB1 interactions with other co-chaperones play a crucial part for folding of the newly generated proteins or in stabilizing and refolding denatured proteins following stress, but, pathologically, is involved in tumorigenesis. For instance, within osteosarcoma, hsa-miR-485-5p binds to the 3'

-untranslated region (UTR) of HSP90 messenger RNA (mRNA) to reduce HSP90 protein production, hence exerting a tumor suppressor effect. Therefore, research is warranted to determine the clinical significance of the lncRNA NNT-AS1/hsa-miR-485-5p/HSP90 axis in CRC patients.

The current study will compare the blood expression level of lncRNA NNT-AS1 and hsa-miR-485-5p, as well as HSP90 serum levels in both healthy and CRC Egyptian patients' cohort peripheral blood samples. Second, examine if lncRNA NNT-AS1/hsa-miR-485-5p/HSP90 axis, or individually investigated, would be used as non-invasive molecular precision biomarker in liquid biopsy for better diagnostic utility for CRC patients. Also, based on CRC patients' group stratification by histologic grades 1-3. Finally, investigate the probable link/correlation between lncRNA NNT-AS1/hsa-miR-485-5p/HSP90 as an axis or individually in CRC Egyptian patients' cohort in relation to demographic data or clinicopathological characteristics. All findings will be confirmed or ruled out by in silico means as well.

3.1. Patient group A total of 60 CRC patients' were enrolled in the study. CRC patients' were treatment-naïve Egyptian patients' cohort admitted to the Clinical Oncology Clinic, National Cancer Institute (NCI), Cairo University, Cairo, Egypt. Male-to-female 1:1 (30/30) and their age range 24-76 years.

3.2. Control group 28 age-matched and sex-matched apparently healthy volunteers, randomly selected from subjects enlisted during normal check-up examination or during blood donation. The control group participants were not taking any medication or suffering from any disease. Controls age range is 40-60 years and 13:15 male-to-female. For the patients group (n = 60) a full history was recorded. If a patient met the inclusion criteria and, after giving their approval for participation in the study and signing the informed consent, peripheral blood samples were taken at the diagnosis time. If a patient met the exclusion criteria, blood samples were not taken. Patient inclusion criteria were those who visited the Colonoscopy Unit for colorectal examination and had a variety of colonic symptoms, including CRC noticeable symptoms, constipation, abdominal pain, rectal bleeding, and sudden weight loss. CRC diagnosis was clinically confirmed by colonoscopy, abdominal radio-imaging, and histopathological examination. Patients exclusion criteria included individuals receiving chemotherapy, radiation, or undergone surgery, patients with blood disorders or any cancer other than CRC. Individuals with inadequate data or missing histopathological diagnoses, as well as those with distant metastases, were excluded from the study.

3.2.1. Patients Pathological and Clinical Data The clinical assessment of CRC patients tumor was done at the Pathology Unit, NCI, Cairo, Cairo University. In addition to a patients colorectal surgery history, the complete family history of cancer disease was recorded for all CRC participants. At the NCI, CRC staging was determined by the colonoscopic results, abdominal radiography, pathological analyses, and clinical decisions, relying on these results and the American Joint Committee on Cancer (AJCC) criteria 2010. Patients are categorized into three stages; stage I/II: local cancer, stage III: lymph node (LN) localized involvement (N1-x), and stage IV: distant metastasis (M1). LN involvement with enlargement incidence as either no (N0) or present (N1), was noted from patient files. The CRC patients family history, smoking status, the noncommunicable diseases status as diabetes mellitus (DM) and hypertension (HTN) were recorded. Tumor site, tumor size, mucinous or not, lymph node metastasis (LNM), tumor invasion or vascular invasion, tumor differentiation, tumor grade, tumor-node-metastasis (TNM) staging, inflammation status as inflammatory bowel disease (IBD), CRC location if colonic or rectal, as well as if transverse, sigmoid, rectosigmoid, and rectal, CRC clinical symptoms, were assessed by the NCI Biochemical Analysis Unit or the Statistics Unit, collected from patients files. Hemoglobin (Hgb), prothrombin time (PT), erythrocyte sedimentation rate (ESR), platelet count, lymphocyte count, lactate dehydrogenase (LDH), C-reactive protein (CRP), were all recorded from patient files done at the NCI, Cairo Egypt, Central Clinical Biochemistry Lab. 4.2. Blood samples Five milliliters of peripheral venous blood liquid biopsy were collected from the antecubital vein from controls and CRC patients into clot activator polymer gel vacutainers. Vacutainers of completely coagulated samples were centrifuged at 4000 r.p.m for 10 min at room temperature (25 ◦C). The collected serum was aliquoted and kept at - 80 ◦C in three DNase/ RNase free Eppendorf tubes until analysis.

4.3. Total RNA extraction Total RNA was extracted from serum samples according to the procedure guidelines. The extracted RNA was dissolved in 40 µL RNase free water and stored in aliquots at - 80 ◦C.

4.4. Quantitation of purified RNA including miRNAs The extracted RNA's purity and concentration are assessed using a spectrophotometer . The quantity of RNA in the sample was assessed using absorbance at 260 nm (A260 = 1 → 44 ng/µL), and RNA purity was assessed using absorbance at 260/280 nm ratios.

4.5. Reverse transcription and expression measurement of ncRNAs using quantitative real-time reverse transcription polymerase chain reaction (qRT-PCR) 4.5.1. lncRNA NNT-AS1 The real-time (RT2) First Strand Kit was used for complementary DNA (cDNA) synthesis as directed by the manufacturer's instructions. The obtained cDNA was stored at - 20 ◦C. After reverse transcription, qRT-PCR was utilized to measure the expression of the lncRNA NNT-AS1 to evaluate the expression level of the lncRNA NNT-AS1, the primer RT2 lncRNA qPCR Assay for Human NNT-AS1 (LPH15988A-200, Cat. No. 330701) was used, and data were normalized using RT2 lncRNA qPCR Assay for Human GAPDH (LPH31725A-200, Cat. No. 330701) as endogenous control. 4.5.2. hsa-miR-485-5p cDNA synthesis was performed as directed by the procedure guidelines. The obtained cDNA was stored at - 20 ◦C. After reverse transcription, qRT-PCR was utilized to measure the expression of the hsa-miR-485-5p. To detect the expression level of the hsa-miR-485-5p, the primer hsa-hsa-miR-485-5p was used and data were normalized miRNA PCR Assay (YP00203901, Cat. No. 339306) as endogenous control. The ncRNA expression level as fold change was calculated and normalized by using the cycle threshold (Ct) approach as fold change (2- ΔΔCt) with GAPDH or SNORD38B (hsa) as the housekeeping genes for lncRNA NNT-AS1 and hsa-miR-485-5p, respectively. ΔCt was calculated by deducting the Ct values of GAPDH and SNORD38B (hsa) from the ones of the lncRNA NNT-AS1 and hsa-miR-485-5p under study, respectively.

ΔΔCt = ΔCt cancer samples - ΔCt control samples where (ΔCt=Ct target - Ct reference) 4.5.3. HSP90 protein quantification by Enzyme-linked immunosorbent assay (ELISA) The HSP90 was quantified by ELISA using the commercially available kit according to the manufacturer's instructions. The Human HSP90 alpha solid-phase sandwich ELISA measures the amount of target bound between a matching antibody pair. In the wells of the supplied microplate, a target-specific antibody has been pre-coated. In these wells, samples, standards, or controls bind to the immobilized (capture) antibody. The sandwich is constructed by adding the second (detector) antibody, followed by the addition of a substrate solution that interacts with the enzyme-antibody-target combination to give a quantifiable signal. This signal's strength is proportional to the concentration of the target in the original material.

4.5.4. CEA and CA19-9 measurement by electrochemiluminescence immunoassay CA19-9 and CEA serum concentrations were measured using an electrochemiluminescence immunoassay using Cobas® e 602, RocheDiagnostics, North America.

4.5.4.1. Routine biochemical testing. Liver function tests: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and serum albumin. Kidney function indicators serum creatinine and urea were determined for all participants.

4.5.5. Ratios and indices Body mass index (BMI) calculation in kg/m2 was done for all the participants, where normal weight = 18.5-24.9 kg/m2 , overweight = 25-29.9 kg/m2 , and obesity = BMI of 30 kg/m2 or greater morbid obesity. Platelet-to-Lymphocytes ratio (PLR) is an immune response-related indicator and systematic inflammation biomarker, which is superior to the neutrophil-to-lymphocytes ratio for correlation with inflammatory disease severity.

ELIGIBILITY:
Inclusion Criteria:

* CRC diagnosed patients that is clinically confirmed by colonoscopy, abdominal radio-imaging, and histopathologicaly.

Exclusion Criteria:

* individuals receiving chemotherapy, radiation, or undergone surgery
* patients with blood disorders
* patients with any cancer other than CRC.
* Individuals with inadequate data or missing histopathological diagnoses
* distant metastases

Ages: 24 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3.1. Patients group A total of 60 CRC pateints' were enrolled in the study. CRC pateints' were treatment-naïve Egyptian patients' cohort admitted to the Clinical Oncology Clinic, National Cancer Institute (NCI), Cairo University, Cairo, Egypt. Male-to-female 1:1 (30/30) and their age range 24-76 years.
  3.2. Control group 28 age-matched and sex-matched apparently healthy volunteers, randomly selected from subjects enlisted during normal check-up examination or during blood donation. The control group participants were not taking any medication or suffering from any disease. Controls age range is 40-60 years and 13:15 male-to-female.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
determination ofncRNA Expression pattern in CRC patients' in comparison to the control group | 9 months
determination of HSP90 protein concentration in control and CRC cases | 12 months
assigning Correlation coefficient between ncRNA, HSP90 protein, CEA, and CA19-9 | 10 months
carry out hsa-miR-485-5p target analysis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hamdy, PhD, Principal Investigator — Faculty of pharmacy Ain Shams University
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Advanced Biochemistry Research Lab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] El-Sheikh NM, Abulsoud AI, Fawzy A, Wasfey EF, Hamdy NM. LncRNA NNT-AS1/hsa-miR-485-5p/HSP90 axis in-silico and clinical prospect correlated-to histologic grades-based CRC stratification: A step toward ncRNA Precision. Pathol Res Pract. 2023 Jul;247:154570. doi: 10.1016/j.prp.2023.154570. Epub 2023 May 24. PMID 37244051
- See also: Publication — https://pubmed.ncbi.nlm.nih.gov/37244051/